CLINICAL TRIAL: NCT07110727
Title: Impact of Capacity Building of Healthcare Workers on Management of Post-Traumatic Stress Disorder Among Road Traffic Injury Patients in Hospitals in Fako Division, Cameroon
Brief Title: Impact of Capacity Building of Healthcare Workers on Management of Post-Traumatic Stress Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Buea (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); University of California, Los Angeles (Other); University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Ngu Claudia Ngeha, Principal Investigator/ PhD Fellow, University of Buea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2024/2524-04/UB/SG/IRB/FHS; D43TW012186 (NIH)
Record Dates: First submitted 2025-07-20; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Post-traumatic Stress Disorder (PTSD) Among Road Traffic Injury Victims
Keywords: Post-Traumatic Stress Disorder; Capacity Building; Screening; PTSD Management; Healthcare workers; Road Traffic Injury; Prevalence; Associated factors; Cameroon
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Study Design This will be a hospital- and community-based intervention study. It will be a sequential study using mixed methods. The study will employ multistage sampling and also involve intervention consisting of capacity building and a non-randomized trial in which a pre/post quasi-experimental design (QED) without a control group will be used to evaluate the feasibility and effectiveness of the intervention (linkage to psychotherapy) in Fako Division, Cameroon. The aim for the QED is to evaluate the feasibility of linkage to mental health care (psychotherapy) in managing PTSD and improving RTI patients' outcomes, as this is a pilot feasibility study, as this has been proven in different settings to be effective; hence there is no equipoise. As a second intervention, the pre/post QED will evaluate the management of PTSD using psychotherapy among 89 (eighty-nine) RTI patients (intervention group) selected by simple random sampling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PTSD cases followed up in a pre/post quasi study for 6 months and pre/post PTSD scores compared. (Experimental): * Intervention 1: Capacity building of healthcare workers Capacity building of healthcare workers on PTSD management. Pre/post capacity building scores of HCWs will be measured and compared (t-test) to assess change in knowledge and comfort level in PTSD management.
  * Intervention 2: Pre/Post Quasi-Experimental Design (QED) with no control group for RTI victims with PTSD.
  A single-arm study with no control group will be included. Participants (RTI patients) diagnosed with PTSD in the baseline study during the determination of the prevalence of PTSD in the intervention group (Buea Regional Hospital) receive psychotherapy during 6 months of follow-up.
  Psychotherapy sessions will be done every two weeks for 6 months. PTSD score measurement and pre/post PTSD score comparison to evaluate the impact of timely management with psychotherapy of PTSD among RTI patients.
  Conclusion and recommendations on trauma quality care improvement of PTSD among RTI patients in HFs in Fako Division.
  Interventions: Behavioral: Two days, role play, adult interactive capacity building sessions of healthcare workers on PTSD screening and management. Pre/posttest and change in practice in screening will be used for evaluation

INTERVENTIONS:
Behavioral: Two days, role play, adult interactive capacity building sessions of healthcare workers on PTSD screening and management. Pre/posttest and change in practice in screening will be used for evaluation — Intervention
  1. Capacity Building of Healthcare workers on PTSD Management For training, the three purposefully selected health facilities selected for the study were written on small pieces of paper. The papers were twisted and thrown on a table. Then, a child was asked to pick up any paper. The one picked was the intervention health facility (Buea Regional Hospital). Healthcare workers at the BRH who provide care to RTI survivors at risk of PTSD 1 month after RTI from our health units of interest in the BRH, will be selected for training (mostly unit heads and front-line staff in trauma/injury will be trained) in two role-play, adult training, interactive sessions on the screening of PTSD using the DSM-5 tool and on timely management of RTI patients with regard to PTSD, linkage to care to psychotherapists, and referrals. Pre/post knowledge evaluation on the use of the DSM-5 tool and management of PTSD will be done, and results compared.

SUMMARY:
This is a community- and hospital-based interventional study consisting of two interventions:

* Capacity building of healthcare workers (HCWs) in the intervention group (Buea Regional Hospital, selected by simple random sampling-balloting method) on management of post-traumatic stress disorder (PTSD) among road traffic injury (RTI) patients (victims). This intervention will be evaluated using pre/posttest scores via a questionnaire to be administered to HCWs to assess change in knowledge and comfort level in PTSD management and 6 months of follow-up to assess change in practice (number of RTI patients screened for PTSD and number of identified PTSD cases referred for treatment to mental health specialists) after the capacity building.
* Also, a pre/post quasi-experimental study design without a control group where psychotherapy will be used in a 6-month follow-up of RTI patients diagnosed with PTSD. The participants (RTI patients diagnosed with PTSD) that will be used for this pre/post quasi-experimental study using psychotherapy will come from the baseline study where the prevalence of PTSD among RTI victims will be determined.

The goal of this clinical trial is to learn if capacity building of healthcare workers on the management (screening, treatment, and referral) of post-traumatic stress disorder (PTSD) among road traffic injury (RTI) patients in hospitals leads to change in knowledge and comfort level of healthcare workers in screening and timely management of PTSD to improve patients' outcomes. Given that attention to care for RTI victims in hospitals in Cameroon and Fako Division in particular is focused on physical care, this study seeks to ensure the provision of holistic care to RTI victims in hospitals, which is in line with the definition of health (comprising the mental, physical, and social well-being of individuals and not just the mere absence of disease or infirmity) by the World Health Organization (WHO). This study will also, through the pre/post quasi-experiment without a control group, learn about the feasibility of using/integrating psychotherapy alongside timely screening for PTSD in routine RTI patient care in primary health care to improve PTSD status in adult RTI patients diagnosed with PTSD in the Cameroonian context.

This study aims to answer five research questions:

Research Questions

1. What is the epidemiological profile of RTI patients at health facilities in Fako Division from 2019 to 2023?
2. What is the prevalence of PTSD among RTI patients in health facilities in Fako Division?
3. What factors are associated with PTSD among RTI patients in health facilities in Fako Division?
4. What is the standard of PTSD care provided to RTI patients in health facilities in Fako Division?
5. What is the impact of capacity building of healthcare workers on the management of PTSD in RTI patients in health facilities in Fako Division? Researchers will

   * Describe the epidemiological profile of RTI patients in hospitals in Fako Division, Cameroon, from January 2019 to December 2023, particularly with regard to PTSD screening recommendation and uptake via an exhaustive chart review of medical records.
   * Determine the prevalence of PTSD among RTI patients via survey using PCL-5 and a cut-off score of at least 33/80.
   * Assess factors associated with PTSD.
   * Assess care given to RTI patients and identify barriers, particularly regarding PTSD management.
   * Compare pre/posttest scores (at baseline-T0, post-training-T1, and 30 days post-training-T2) of healthcare workers' knowledge and comfort level in PTSD management following capacity building of HCWs on PTSD management to see if there is change in knowledge and comfort level due to the capacity-building intervention in the randomly selected hospital chosen as the intervention group (Buea Regional Hospital) and also establish if the knowledge was sustained after 30 days.
   * Collect data at 1, 3, and 6 months of follow-up on the number of RTI patients screened for PTSD by trained health workers during 6 months of post-training follow-up and the number of timely referrals of PTSD cases identified, and compare these to what was obtained before the training (baseline) and establish if there is a change.
   * Collect data on the PTSD status of PTSD patients at 1, 3, and 6 months of follow-up with psychotherapy and conclude on the feasibility of including psychotherapy in the Cameroonian context to improve PTSD status.

Participants (RTI victims) will:

* Be booked for PTSD screening 1 month after RTI, be called up for an appointment to be screened 1 month after RTI, and have diagnosed PTSD cases referred for effective management.
* Diagnosed PTSD cases will be followed up with psychotherapy once every 2 weeks for 6 months (12 sessions in total), and PTSD status will be followed up monthly.
* Keep a record of symptoms, difficulties/challenges faced in managing PTSD, the number of times they experience PTSD symptoms, and improvement over time.

DETAILED DESCRIPTION:
Abstract Background: Road traffic injuries (RTIs) are a major global public health concern, often leading to serious physical and psychological consequences, including post-traumatic stress disorder (PTSD), a prevalent and debilitating psychiatric disorder following RTIs. About 22.2% of RTI victims develop PTSD worldwide and several factors have been associated with PTSD in RTI. Victims of RTIs frequently present to primary care, however PTSD in RTI patients remain under-explored in low and middle income (LMIC) settings like Cameroon and there is no standardized practice on the routine screening of PTSD among RTI. Late identification of PTSD and/or poor management could become fatal to health system. Timely management is the most viable way of closing the gap. Objectives: Study aims to evaluate the impact of capacity building of Health care workers on management of PTSD among RTI patients in Health Facilities (HFs) in Fako. Materials and methods: A hospital and community-based intervention study will be conducted at three purposefully selected hospitals in Fako Division, Cameroon: Buea Regional Hospital, Saint Luke Hospital Buea, and Limbe Regional Hospital. These hospitals are selected because of the frequency of RTI patients visiting the hospitals. Buea Regional Hospital was selected as the intervention group via simple random sampling. Using a sequential design, the study included; a hospital chart review aimed at establishing the epidemiological profile of RTI over 5 years (2019-2023), cross sectional study aimed at determining the prevalence and factors associated with PTSD (January 2023 to June 2024), and exploratory study (in-depth interviews and cross sectional study) aimed at assessing care given to RTI patients and identify gaps in PTSD care and barriers to PTSD management. The intervention will consist of capacity building of healthcare workers on management of PTSD in RTI victims with pre/posttest used for evaluation, and the use of psychotherapy in a pre/post quasi experimental study without a control group for 89 selected patients that will be diagnosed with PTSD aimed at improving patients' outcome (PTSD score/status). Consenting adult RTI survivors, aged 18years and above will be recruited and standardized DSM-5 PTSD checklist will be used for PTSD diagnosis. Qualitative data will be analyzed using thematic approach and quantitative data inputted into kobo toolbox and analyzed in SPSS using descriptive statistics and binary logistic regression at 5% level of significance. Expected outcomes: Consist of the epidemiological profile of RTI patients, RTI trends over 5years, prevalence and factors associated with PTSD in RTI, standard of care given to RTI patients particularly regarding PTSD care in RTI victims by HCWs, barriers to PTSD management. The impact of capacity building of HCWs on PTSD management; change in knowledge and comfort level in PTSD screening, and management by HCWs. Number of RTI patients screened for PTSD by trained HCWs during 6 months post-training follow-up, number of timely referrals of PTSD cases identified, and PTSD patients' PTSD score/status (outcomes) at 1,3,and 6 months follow-up with psychotherapy. This study will improve patients' outcomes and provide evidence for in-hospital care quality improvement, inform policy and practice.

INTRODUCTION 1.1 Background to the Study Post-traumatic stress disorder (PTSD), a serious mental health condition triggered by traumatic events such as road traffic injuries (RTIs), represents a significant yet often overlooked consequence of RTIs, adding a substantial mental health burden to the already significant physical trauma. While RTIs are recognized as a major global public health challenge, the psychological impact on survivors, particularly the development of PTSD, often remains underreported and undertreated, especially in low- and middle-income countries (LMICs) like Cameroon. To address this critical gap in care, there is a pressing need to build the capacity of healthcare workers (HCWs) in Fako Division- Cameroon to effectively screen for, diagnose, and manage PTSD among RTI patients, thereby facilitating holistic recovery and improving patients' outcomes.

Road traffic Injuries are a significant global public health problem and a leading cause of morbidity, mortality, and disability, disproportionately affecting low- and middle-income countries (LMICs) where over 93% of the world's RTI-related fatalities occur. Organized trauma care systems have been shown to save lives and reduce morbidity. Globally, RTIs result in about 1.35 million deaths annually, with 20-50 million sustaining severe injuries. Reports from WHO in 2022 indicate that road traffic crashes (RTCs) cost most countries 3% of the gross domestic product (GDP), with the highest rates of RTI recorded in the African region.

Beyond the fatal consequences, RTIs also cause significant morbidity with social, professional, economic, physical, and psychological consequences, with post-traumatic stress disorder (PTSD) being a prevalent and debilitating mental health issues. Road traffic injury (RTI) is one of the principal causes of PTSD, ranking third after sexual and physical assaults. The World Health Organization (WHO) recognizes mental health as an integral component of overall well-being, and has identified PTSD as a significant public health concern, including PTSD in the priority conditions covered by WHO's mental health Gap Action Programme (mhGAP), which includes guidelines for managing PTSD, emphasizing the need for comprehensive care, especially in LMICs. PTSD is diagnosed using the PTSD checklist-5 (DSM-5) and is characterized by intrusive recollections, avoidance behaviors, negative alterations in cognition and mood, and hyper arousal, which can profoundly impair an individual's ability to function, reintegrate into society, and lead a fulfilling life.

Studies consistently demonstrate a significant prevalence of PTSD among RTI survivors globally. Recent meta-analysis and systematic review suggests that the global prevalence of PTSD among RTI survivors ranges from 6.3% to 58.3% with a pooled prevalence of 22.2%, varying based on factors such as population characteristics, time elapsed since the injury, and assessment methodologies. Prior research across Africa consistently reveals a substantial burden of PTSD, with pooled prevalence estimates reaching 26% ranging from 8% to over 61%, underscoring the substantial psychological burden associated with RTIs. Untreated PTSD can profoundly impair an individual's ability to function, reintegrate into society, and maintain overall well-being, thereby leading to substantial personal suffering and escalating societal costs. All demographics are indiscriminately affected by PTSD, and several factors have been associated with the development of PTSD in RTI.

In Cameroon, a LMIC, RTIs represent a significant and growing public health concern, ranking as the 8th leading cause of disability-adjusted life years (DALYs), and leading cause of morbidity and mortality. About 16,583 road crashes occur each year, with over 1,000 deaths from government records, and approximately 6000 according to WHO estimates, with the burden reflected in the estimated 1443 disability-adjusted life years (DALYs) per 100,000 population lost to road crashes. Several factors contribute to the high incidence of RTIs, including rapid urbanization, poor road infrastructure, inadequate enforcement of traffic laws, and the widespread use of motorcycles as an affordable mode of transportation. In the South West Region, the presence of socio-political crises has further amplified the risk of RTIs, specifically in the Fako Division, with internally displaced persons (IDPs) increasingly relying on motorcycles for livelihoods, predisposing them to RTI. While the Cameroonian government has undertaken commendable efforts to improve road safety through awareness campaigns and infrastructure development projects, the psychological consequences of RTIs have often received insufficient attention. Cameroon has integrated mental health into its minimum package of healthcare services, aligning with WHO recommendations, however, routine screening for prevalent mental health disorders like PTSD is not yet standard practice in primary healthcare. Moreover, specialized mental health resources, including psychiatrists, are disproportionately concentrated in major cities such as Douala and Yaounde, limiting access in areas like the Fako Division. The interplay between physical injuries and mental health consequences in the aftermath of RTI highlights the holistic impact these incidents have on victims.

Given the circumstances, there is a pressing need to enhance the capacity of healthcare workers (HCWs) in Cameroon, particularly in areas like Fako Division, to provide comprehensive care that addresses both the physical and psychological needs of RTI survivors. Equipping HCWs with the necessary knowledge, skills, and evidence-based practices for early PTSD detection and management holds the potential to improve patients' outcomes, enhance quality of life, and mitigate the long-term consequences of RTIs. Studies demonstrate that early screening improves both patient care and outcomes for trauma victims. Various intervention models, including the Donabedian's Structure-Process-Outcome model and the stepped-care model have been used to improve practice in healthcare.

1.2 Statement of the Problem Despite the World Health Organization's (WHO) recognition of mental health as an integral component of overall well-being (WHO), and the integration of mental health services into Cameroon's minimum healthcare package, the mental health needs of road traffic injury (RTI) survivors in Fako Division remain largely unmet. While physical injuries caused by RTIs receive quick attention and treatment, psychological repercussions, notably the development of post-traumatic stress disorder (PTSD), are often overlooked or inadequately addressed. This neglect stems from a complex interplay of factors, including limited awareness among healthcare providers, a shortage of trained mental health professionals, a lack of standardized screening protocols, and widespread stigma around mental illness.

Despite the well-documented link between RTIs and PTSD, as well as the disproportionate impact of RTIs, especially in LMICs, with one in four RTI survivors in Africa experiencing PTSD. PTSD in RTI remains under-resourced and under-prioritized in Cameroon, where routine screening for PTSD is lacking in primary care for RTI victims. This screening gap represents a considerable barrier to early detection and management. Even when PTSD is suspected, access to specialized mental health services is severely limited as the majority of psychiatrists and psychologists are concentrated in major urban centers such as Douala and Yaoundé, leaving areas like Fako Division with few, if any, mental health specialists. This geographical disparity in access to care creates a significant challenge for RTI survivors who require specialized psychological treatment.

Furthermore, few trauma centers and hospitals monitor and address mental health recovery in low and middle-income (LMIC) countries such as Cameroon with frequent oversight of Post-Traumatic Stress Disorder (PTSD), a prevalent mental health condition after RTI. This can severely compromise the recovery and overall well-being of victims. This oversight is particularly concerning in LMICs like Cameroon, where limited resources and competing health priorities often overshadow mental health needs. This deprives patients of achieving holistic health, encompassing mental, physical, and social well-being, beyond the mere absence of disease as defined by WHO.

The absence of PTSD data in the Cameroon Trauma Registry (CTR) limits policy, guidelines, and interventions targeting this critical public health issue. In Fako Division, Cameroon, RTI is a significant public health concern, imparting physical and psychological burdens on survivors that often manifest as PTSD. Injury in the South West region of Cameroon is associated with significant disability and lost productivity. Injury-related mortality in this region is estimated to be 113 per 100,000 person-years, exceeding estimated Cameroonian death rates for malaria and tuberculosis combined. Poor management of trauma/injury may lead to poor trauma outcomes, including PTSD. Primary healthcare facilities are typically the first point of contact for RTI victims seeking medical assistance, however PTSD screening is not integrated into routine primary healthcare checks after RTCs in Fako Division. This underscores the need for comprehensive care, including mental health support, to address the holistic needs of RTI survivors.

Despite the substantial burden of RTIs in Cameroon there is a paucity of data on RTIs, particularly about PTSD screening uptake in RTI in Cameroon. Hence, limiting the understanding of specific RTI patient characteristics, particularly regarding PTSD screening recommendation and uptake in Cameroon. Within Cameroon, data on the epidemiological characteristics of RTI patients and associated mental health conditions such as PTSD remain scarce, especially at the sub-national level, with previous research focusing only on RTI patients' demographic and injury characteristics.

This issue is further exacerbated by a paucity of data on the prevalence and factors associated with PTSD among RTI patients in the country, as previous research has mainly concentrated on PTSD in the contexts of HIV/AIDS and conflict. Late identification of cases and/ or poor management of this condition could become fatal to the health system; increasing health costs, increasing healthcare utilization, and increasing the National burden financially and otherwise (productivity of the victim and family members affected). PTSD not only affects those who suffer from the illness, but also extends and affects the communities in which crisis intervention is not regularly implemented.

The care delivered to RTI patients with PTSD in Fako remains uncertain, necessitating an assessment to identify care gaps to enhance service delivery and ensure patient-centric care models align with best practices and evidence-based standards. In addition, the limited capacity among healthcare workers (HCWs) in managing PTSD among RTI patients exacerbates the issue. HCWs require training and support to be effective in screening for and managing PTSD in RTI survivors. The lack of standardized guidelines and protocols for PTSD management in hospitals in Cameroon further compounds the problem. To reduce avoidable morbidity and, in extreme situations, death from injury, all links in the chain of survival after RTC need strengthening to close the gap. Addressing both the physical and mental well-being of individuals affected by RTI in hospitals is crucial for comprehensive care and optimal recovery. Given its significant impact on individuals, the economy, and the health system, routine screening for PTSD in suitable settings is crucial.

The consequences of untreated PTSD can be severe and long-lasting, affecting not only the individual but also the families, communities, and nations. PTSD can lead to lower health-related quality of life, higher rates of physical health symptoms, and increased risk for premature mortality. Comorbidity is prevalent, with 80-90% of PTSD patients having one or more additional diagnoses, commonly major depression, anxiety disorders, substance use disorders, borderline personality disorder, and psychotic disorders. In addition, some patients show additional symptomatic features such as suicidal ideation, dissociation, physical health problems, limited work and social functioning, difficulties finding work, divorce, and violence, which may affect 84% of people with PTSD making things more difficult. Many trauma patients report emotional or psychological distress after injury (19-42%), and this is associated with deficits in physical recovery, social functioning, and quality of life.

Furthermore, PTSD can have far-reaching consequences, including obesity, pain, cardiovascular diseases, diabetes, hypertension, impairment, and difficulties in recovery and treatment. Not screening for PTSD can lead to an incorrect diagnosis and inappropriate treatment, which in turn can lead to permanent damage and life-threatening behaviors. Given that comorbidity is the norm rather than the exception among PTSD patients, and the potential for incorrect diagnoses and inappropriate treatment due to lack of screening, an important question to answer is, whether primary health care providers in Cameroon and Fako Division in particular who are the first point of contact for care to majority of RTI victims are capacitated to; identify, screen and timely manage PTSD among RTI patients to improve patients outcome and wellbeing.

Despite the prevalence of PTSD in RTI victims in the literature, consequences and associated comorbidities, a comprehensive understanding of the epidemiology, prevalence, associated factors, and care standards concerning PTSD remains elusive among RTI victims in Fako specifically and Cameroon in general. The absence of such data hampers tailored interventions, widens gaps in mental health support, and hinders optimal care delivery to RTI patients grappling with PTSD at health facilities in Fako Division. This highlights the urgent need for PTSD capacity-building initiatives targeting HCWs to enhance PTSD management practices to mitigate the psychological impacts of RTI/trauma in this population.

1.3 Justification for the Study This study addresses the pressing need to improve mental health support for RTI patients in Fako Division, Cameroon. RTIs inflict not only physical harm but also enduring mental health consequences, with post-traumatic stress disorder (PTSD) emerging as a prevalent and debilitating consequence. The World Health Organization (WHO) recognizes PTSD as a significant public health concern, including PTSD in the priority conditions covered by WHO's mental health Gap Action Programme (mhGAP), which includes guidelines for managing PTSD, emphasizing the need for comprehensive care, especially in LMICs.

Despite these global efforts, a lack of comprehensive understanding of the burden of PTSD in RTI (prevalence and associated factors), care gaps in PTSD management for RTI victims, and the impact of tailored interventions and capacity-building initiatives for HCWs are lacking in Fako Division and Cameroon at large. This exacerbates the suffering of RTI survivors, impeding recovery and perpetuating long-term societal burdens. The absence of routine screening and inadequate care for PTSD among RTI patients in Cameroon underscores the urgency of this research, which aims to fill these knowledge and practice gaps, drive evidence-based interventions, and inform policy recommendations tailored to the unique needs of RTI patients in Fako and similar settings.

This study's evaluation of HCWs' capacity in PTSD management, as well as its goal of closing the gap by building capacity for identifying, screening, and referring/treating PTSD, will help to improve mental health care, improve patient outcomes, and reduce the burden of PTSD on individuals, families, and communities. The findings will help inform healthcare practices, policy development, and patient care, reducing the long-term impact of RTIs on mental health and promoting resilient and sustainable health systems.

This research is consistent with global health goals, notably Sustainable Development Goal (SDG) 3, which emphasizes healthy lives and well-being for all ages. This study contributes to the long-term development of tailored mental health interventions in low- and middle-income countries by improving trauma care quality for RTI patients in Fako Division through the implementation of evidence-based screening protocols, capacity-building initiatives, and quality enhancement efforts.

There is limited existing research and a paucity of data on PTSD among RTI patients in Cameroon. The findings of this study will provide insights into the epidemiological profile of RTI patients in Fako, Cameroon, with a focus on PTSD screening practices, prevalence rates, risk factors, and care gaps; information critical to informing targeted interventions and policy recommendations. It will provide data based on local evidence to advocate for the integration of systematic screening and timely treatment of PTSD into the routine management of RTI patients in Cameroon and similar LMIC settings, since early diagnosis and management are critical to improving patient outcomes.

Ultimately, this research seeks to contribute to a more holistic and equitable approach to RTI care in hospitals, one that acknowledges and addresses the frequently overlooked psychological needs of RTIs survivors. This research has the potential to drive transformative change in healthcare practices, policy development, and patient outcomes, improving the lives of RTI survivors and the families in Cameroon.

Data from the Cameroon Trauma Registry (CTR), indicates that RTC accounts for over 60% of all injury presenting to the emergency department of the Limbe regional hospital, in Fako Division. However, the extent to which victims are psychologically affected is not well known. To the best of our knowledge, no study has been carried out to determine the prevalence or risk factors of PTSD in RTI. Given the public health importance and burden from the literature, it is important to carry out this study as a pilot study to determine this burden and evaluate the impact of capacity building of health care workers on PTSD management as an intervention to improve patient outcomes. This study has the potential to provide data based on local evidence to inform the improvement of the quality of care to RTI patients with PTSD, necessary to inform practice and policy.

Studies have shown that early interventions for PTSD, such as screening, can improve patient outcomes and overall quality of life, and recommend that further studies are needed. No intervention for PTSD in RTI victims has been carried out in Cameroon using the education of HCWs. Investigators aim to carryout this pilot intervention study to evaluate the impact of capacity building of HCWs on PTSD management of RTI victims. Early screening is crucial to identify cases which otherwise will be missed or overlooked.

This research is essential to bridging knowledge gaps, improving clinical practice and patient outcomes, and inform policy. It will be important and instrumental in the way health services assess and treat RTI/trauma victims presenting in HFs with mental health problems like PTSD, will reduce burden of PTSD both emotionally and financially at individual, community and national levels.

1.4 Research Hypotheses Investigators hypothesize;

1. Motorbike riders are the most involved in RTI over the last five years in Fako.
2. There is a high prevalence of PTSD among RTI survivors in Fako.
3. Post-traumatic stress disorder is associated with duration since RTI.
4. Inadequate care; absence of routine screening for PTSD, is given to RTI survivors with PTSD in Health Facilities in Fako.
5. Capacity building of healthcare workers on PTSD screening and management will lead to improved healthcare workers' knowledge and skills, increase the proportion of cases of PTSD that are timely screened and managed, improve quality of PTSD care, and improve patient outcome by reducing symptoms and will lead to reduction of PTSD score in intervention group.

1.5 Research Objective 1.5.1 General Objective The main objective of this study is to evaluate the impact of capacity building of health care workers on the management of Post-Traumatic Stress Disorder among Road Traffic Injury Patients in Health Facilities in Fako Division.

1.5.2 Specific Objectives

1. To describe the epidemiological profile of RTI patients at Health Facilities in Fako Division from 2019 to 2023.
2. To determine the prevalence of PTSD among RTI patients at Health facilities in Fako Division.
3. To assess the factors associated with PTSD among RTI victims in Fako Division.
4. To assess the care given to RTI patients with PTSD and identify PTSD care gaps in Health Facilities in Fako Division.
5. To evaluate the impact of capacity building of healthcare workers on management of PTSD among RTI patients in Fako Division.

1.6 Conceptual Framework for the Study This study's conceptual framework is grounded in Donabedian's Structure-Process-Outcome (SPO) model of healthcare quality, developed in 1966 by Avedis Donabedian. This model provides a framework for examining health services and evaluating quality of health care. The model posits that the quality of care is determined by three interconnected elements: structure, process, and outcome. Donabedian argued that improvements in the structure of care should lead to improvements in clinical processes, which, in turn, should result in improved patient outcomes. "Process" is defined as the sum of all actions that make up healthcare done to and for the patient (e.g. screening, treatment, preventive care, and patient education, referrals,); "outcome" contains all the effects of healthcare on patients or populations (e.g., changes to health status, behavior, or knowledge as well as patient satisfaction and health-related quality of life); and "structure" includes all of the factors that affect the context in which care is delivered. (e.g., screening tools/equipment, availability of psychotherapy, physical facility, equipment, and human resources, as well as organizational characteristics such as staff training and payment methods) This study adapts the features of this model to develop a framework for evaluating the impact of capacity building of HCWs on PTSD management and the subsequent improvement in PTSD outcomes among RTI victims in hospitals in Fako Division. This study illustrates the relationship between the capacity building (intervention) of HCWs (a structural component focused on healthcare worker training) and the management of PTSD (a process component encompassing screening, treatment, referral, and supervision), ultimately influencing PTSD outcomes (the outcome component reflecting PTSD status) among road traffic injury (RTI) patients. The interplay between different processes are crucial for effective PTSD management and improved outcomes, 1.7 Study Duration The study will last 15 months; from July 2024 to September 2025 and will consists of four phases.

* Phase 1- the pre-intervention phase (In-depth interview, cross sectional study); will consist; chart review, exploratory (in-depth interview (IDI) and cross sectional) study for 2 months. This will be carried out in all the 3 selected health facilities (HFs). In-depth interview will be conducted with HF administrators and/ unit heads (in units involved with RTI victims care) using in-depth interview guide to capture quality of care and identify gaps for HCWs capacity building. Baseline data will be collected from July 2024 to December 2024 by direct administration of pretested structured questionnaires to patients and HCWs as necessary. Medical records review (from registers at the different units involved with RTI patient care) will also be used to collect baseline medical data of RTI survivors.
* Phase 2 (Intervention); this will consist of the intervention which involves 2 sessions of capacity building of health care workers involved in RTI patients' care in our units of interest in the Buea Regional hospital which was selected as intervention site by simple random sampling (balloting method).
* Phase 3- post intervention (Pre/post Quasi experimental design, QED without a control group will last 6 months (QED) and starts after capacity building of HCWs on PTSD management. After building the capacity of HCWs on PTSD screening and management. PTSD cases diagnosed at the BRH (by researchers when determining PTSD prevalence) will be selected for intervention using simple random sampling. A pre/post quasi experiment without a control group will be used where the patients will be followed-up with psychotherapy for 6 months. PTSD scores will be measured at time intervals at; 1, 3 and 6 months. Pre/post comparisons of the different data will be done to evaluate the impact of capacity building and management (PTSD screening and referral to psychotherapy) of PTSD in RTI patients in the HFs.

A) Exploratory Sequential exploratory mixed-methods design made up of qualitative and quantitative methods will be used. The exploratory study will start with the qualitative method (in-depth interview), then end with the quantitative method (questionnaire). The intervention consist of capacity building of HCWs on screening and management of PTSD and thereafter the use of a pre/post quasi experimental study design (with no control) using psychotherapy as a feasibility study.

B) Interventions and Random Allocation

* Intervention 1; Capacity building of HCWs on screening and PSTD management. This will be a hospital-based capacity building of Healthcare workers from the Buea Regional Hospital (BRH) and will be done at the BRH. A pre/posttest will be used for evaluation. Healthcare workers/ staff at the BRH, who provide care (general screening, diagnosis and treatment) for RTI survivors at risk for PTSD one month after survival period will be trained. Currently in the BRH, PTSD screening is not part of routine screening at HFs in Fako. While training and education will be focused on this group, other providers/ staff will be welcomed to attend the capacity building sessions. The level of training for this is universal and does not depend on the trainees' background (Medical Doctor/ nurse). This study is a feasibility pilot study with goal to get people screen for PTSD and linkage to care. A training manual will be used with the intervention package consisting; a 2 day on site interactive training sessions using adult training method including role play for skills building, provision of educational materials, resources (DSM-5 for screening and psychotherapist for linkage to care), supervision and collaboration. A pre/post evaluation will be done to evaluate our intervention (capacity building). A predesigned training manual by the principal investigator and facilitators (clinical psychologist/mental health expert) will be used. Role play will be done to facilitate mastery of the training received with questions and answer sessions done using an interactive approach. The training will end with a posttest questionnaire to evaluate capacity building of the HCWs (pre/post test results comparison using t-test) and follow-up post training evaluation at 1,3 and 6 months.
* Intervention 2; Pre/ Post Quasi Experimental study design without control This study employs a pre/post quasi-experimental design to evaluate the effectiveness and feasibility in the Cameroonian context the use of psychotherapy in reducing symptoms of PTSD) among RTI patients. The study will be conducted at the Buea Regional Hospital (BRH), which was selected via simple random sampling from three hospitals: BRH, Saint Luke Hospital (SLH), and Limbe Regional Hospital (LRH). RTI patients who were diagnosed with PTSD during the baseline data collection will be eligible for the psychotherapy intervention. A total of about 89 PTSD-positive patients will be randomly selected from the BRH site using a simple random sampling technique.

The psychotherapy intervention will consist of two sessions per month for 6 months , each session lasting about 60 minutes conducted by trained psychotherapists using a standardized protocol. Evaluation of psychotherapy intervention will be done by comparing the pre/post PTSD score/status.

ELIGIBILITY:
Inclusion criteria for healthcare workers for capacity building:

* Health care workers at the selected hospital for intervention in Fako Division (Buea Regional Hospital).
* Involved in trauma/RTI injury care.
* Have at least one year of working experience with RTI patients.
* At least 18 years old and above and consent to the study.

Exclusion criteria:

- Healthcare worker who will be sick or not available on days of the training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible RTI survivors screened for PTSD at the 1-month follow-up visit in the hospital. | Measured at 1 month post-injury (following capacity building of HCWs) and followed up for 6 months.
  The percentage of eligible road traffic injury (RTI) survivors presenting to the participating health facility for the intervention (Buea Regional Hospital) who are screened for Post-Traumatic Stress Disorder (PTSD) using a standardized screening tool (e.g., PCL-5) at the participants (RTI survivors) 1-month follow-up visit following capacity building of healthcare workers. The unit of measurement is percentage.

SECONDARY OUTCOMES:
Change in healthcare workers Knowledge of PTSD management. | Day 1 (baseline), day 2 (at the end of training), and day 30 (after capacity building).
  Improvement in healthcare workers (HCWs) knowledge scores (based on a structured questionnaire) regarding PTSD management in road traffic injury victims.
Change in Healthcare worker Comfort (HCW) Level in PTSD Management | Day 1 (baseline), day 2 (at the end of training), and day 30 (after the capacity-building intervention).
  Improvement in self-reported comfort level scores (based on a structured questionnaire) about HCWs level of comfort regarding PTSD management, measured at day 1 (baseline), day 2 (end of training), and 30 days after training.
Proportion of PTSD-positive screens referred for treatment. | 6 months after training
  The percentage of RTI survivors who screen positive for PTSD and are subsequently referred for mental health treatment by trained HCWs. This will be monitored for 6 months after training of HCWs.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Ngeha Ngu, PhD Fellow, Principal Investigator — University of Buea
Locations (3):
- Cameroon (3):
  - Buea Regional Hospital, Buea
  - Saint Luke Hospital, Buea
  - Limbe Regional Hospital, Limbe

IPD SHARING:
Plan to Share IPD: Yes
Individual participants data that underline the results reported in the study will be made available after de-identification. Data will be shared with researchers who provide methodologically sound proposals and agree to use data only for research purposes. Data will be available starting 6 months after publication and for upto 5 years. To request access, contact the principal investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication and 5 years after the start date
Access Criteria: Individual participant data (IPD) and supporting documents will be accessible to qualified researchers who submit a scientifically sound research proposal related to the study objectives. Researchers must agree to use data solely for research purposes and to maintain participant confidentiality. Access will be granted after approval by the principal investigator or the study steering committee. Data and documents will be shared via secure data transfer methods upon signing a data use agreement. Requests can be submitted by contacting the principal investigator at nguclaudia2018@gmail.com
URL: https://www.ubuea.cm

REFERENCES:
- See also: Preprint of the study on epidemiological profile of road traffic injury patients in hospitals in Fako division, Cameroon: a foundation for tailored post-traumatic stress disorder (PTSD) management. It is available at medRxiv — https://doi.org/10.1101/2025.06.10.25329319